CLINICAL TRIAL: NCT03433248
Title: RACELINES: Renal Actions of Combined Empagliflozin and LINagliptin in Type 2 diabetES
Brief Title: Renal Actions of Combined Empagliflozin and LINagliptin in Type 2 diabetES
Acronym: RACELINES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.H.H. Kramer (Other)
Responsible Party: Sponsor-Investigator, M.H.H. Kramer, Head of the Internal Medicine department, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DC2017RACELINES01
Record Dates: First submitted 2017-11-22; First posted 2018-02-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Type2 Diabetes
Keywords: Type 2 diabetes mellitus; Diabetic kidney disease; Diabetic nephropathy; Renoprotection; SGLT2 inhibitor; Empagliflozin; DPP-4 inhibitor; Linagliptin; SU derivative; Gliclazide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — empagliflozin; Linagliptin; Gliclazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMPA/LINA 10/5 mg QD (n=22) (Experimental): 8w EMPA followed by 8w EMPA/LINA 10/5 mg QD (n=22)
  Interventions: Drug: EMPA/LINA 10/5 mg QD (n=22); Drug: LINA/EMPA 5/10 mg QD (N=22)
- LINA/EMPA 5/10 mg QD (N=22) (Experimental): 8w LINA followed by LINA/EMPA 5/10 mg QD (N=22)
  Interventions: Drug: EMPA/LINA 10/5 mg QD (n=22); Drug: LINA/EMPA 5/10 mg QD (N=22)
- Gliclazide 30 mg QD/BID (N=22) (Active Comparator): 8w Gliclazide 30 mg QD, followed by 8w Gliclazide BID (N=22)
  Interventions: Drug: Gliclazide 30 mg QD/BID (N=22)

INTERVENTIONS:
Drug: EMPA/LINA 10/5 mg QD (n=22) — Once daily treatment with oral empagliflozin (Jardiance) 10 mg Once daily treatment with oral linagliptin (Tradjenta) 5 mg
  Other Names: Jardiance; Tradjenta
  Arms: EMPA/LINA 10/5 mg QD (n=22); LINA/EMPA 5/10 mg QD (N=22)
Drug: LINA/EMPA 5/10 mg QD (N=22) — Once daily treatment with oral linagliptin (Tradjenta) 5 mg Once daily treatment with oral empagliflozin (Jardiance) 10 mg
  Other Names: Tradjenta; Jardiance
  Arms: EMPA/LINA 10/5 mg QD (n=22); LINA/EMPA 5/10 mg QD (N=22)
Drug: Gliclazide 30 mg QD/BID (N=22) — Once daily or twice daily treatment with oral glicazide MR 30mg
  Other Names: Gliclazide Sandoz
  Arms: Gliclazide 30 mg QD/BID (N=22)

SUMMARY:
The current study aims to explore the clinical effects and mechanistics of mono- and combination therapy with SGLT-2 inhibitor empagliflozin and DPP-4 inhibitor linagliptin on renal physiology and biomarkers in metformin-treated T2DM patients.

DETAILED DESCRIPTION:
Sodium-glucose linked transporters (SGLT-2) inhibitors and dipeptidyl peptidase-4 (DPP-4) inhibitors are relatively novel glucose-lowering drugs for the treatment of T2DM. These agents seem to exert pleiotropic actions 'beyond glucose control'. SGLT-2 inhibitors decrease proximal sodium reabsorption and decrease glomerular pressure and albuminuria in rodents and type 1 diabetes patients. In addition, SGLT-2 inhibitors reduce, blood pressure and body weight. In rodents, SGLT-2 inhibitors also improved histopathological abnormalities associated with DKD. DPP-4 inhibitors are considered weight neutral, improve lipid profiles and slight reductions in blood pressure have been reported. To date, the potential renoprotective effects and mechanisms of SGLT-2 inhibitors and combination therapy with SGLT-2 inhibitors have not been sufficiently detailed in human type 2 diabetes. The current study aims to explore the clinical effects and mechanistics of mono- and combination therapy with an SGLT-2 inhibitor and a DPP-4 inhibitor on renal physiology and biomarkers in metformin-treated T2DM patients.

66 patients with type 2 diabetes will undergo a 16-week intervention period with 8-week empagliflozin (SGLT-2 inhibitor) monotherapy, followed by 8-week empagliflozin and linagliptin (DPP-4 inhibitor) combination therapy or 8-week linagliptin monotherapy, followed by 8-week linagliptin and empagliflozin combination therapy or 8-week gliclazide (SU derivative), followed by 8-week gliclazide intensification therapy in order to assess changes in the outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian*
* Both genders (females must be post-menopausal; no menses >1 year; in case of doubt, Follicle-Stimulating Hormone (FSH) will be determined with cut-off defined as >31 U/L)
* Age: 35 - 75 years
* BMI: >25 kg/m2
* HbA1c: 7.0 - 9.5% Diabetes Control and Complications Trial (DCCT) or 53 - 80 mmol/mol International Federation of Clinical Chemistry (IFCC)
* Treatment with a stable dose of oral antihyperglycemic agents for at least 3 months prior to inclusion
* Metformin monotherapy
* Combination of metformin and low-dose SU derivative**
* Hypertension should be controlled, i.e. ≤140/90 mmHg, and treated with an ACE-I or ARB (unless prevented by adverse effect) for at least 3 months.
* Albuminuria should be treated with a RAAS-interfering agent (ACE-I or ARB) for at least 3 months.
* Written informed consent

  * In order to increase homogeneity ** In order to accelerate inclusion, patients using combined metformin/SU derivative will be considered. In these patients, a 12 week wash-out period of the SU derivative will be observed, only when combined use has led to a HbA1c <8% at screening. Subsequently, patients will be eligible to enter the study, now using metformin monotherapy, provided that HbA1c still meets inclusion criteria.

Exclusion Criteria:

* Estimated GFR <45 mL/min/1.73m2 (determined by the Modification of Diet in Renal Disease (MDRD) study equation)
* Hemoglobin level < 7.0 mmol/L
* Current urinary tract infection and active nephritis
* History of unstable or rapidly progressing renal disease
* Macroalbuminuria; defined as ACR of >300 mg/g.
* Current/chronic use of the following medication: thiazolidinediones, sulfonylurea derivatives, GLP-1 receptor agonists, DPP-4 inhibitors, SGLT-2 inhibitor, oral glucocorticoids, immune suppressants, antimicrobial agents, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs) and monoamine oxidase inhibitors (MOAIs).
* Patients on diuretics will only be excluded when these drugs cannot be stopped 3 months prior randomization and for the duration of the study.
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications (i.e. sports injury, head-ache or back ache). However, no such drugs can be taken within a time-frame of 2 weeks prior to renal-testing
* Pregnancy
* History of or actual severe mental disease
* History of or actual severe somatic disease (e.g. systemic disease)
* History of or actual malignancy (except basal cell carcinoma)
* History of or actual pancreatic disease
* (Unstable) thyroid disease
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN)
* Recent (<6 months) history of cardiovascular disease, including

  * Acute coronary syndrome
  * Stroke or transient ischemic neurologic disorder or chronic heart failure (NYHA grade II-IV)
* Complaints compatible with or established neurogenic bladder and/or incomplete bladder emptying (as determined by ultrasonic bladder scan)
* Substance abuse (alcohol: defined as >3 units alcohol/day)
* History of diabetic ketoacidosis (DKA) requiring medical intervention (e.g., emergency room visit and/or hospitalization) within 1 month prior to the Screening visit.
* Recent blood donation (< 6 months)
* Allergy to any of the agents used in the study
* Inability to understand the protocol and/or give informed consent
* Individuals who are investigator site personnel, directly affiliated with the study, or are immediate (spouse, parent, child, or sibling, whether biological or legally adopted) family of investigator site personnel directly affiliated with the study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
GFR | 16 weeks
  Changes from baseline following 16-week treatment on renal hemodynamics in both the fasting and postprandial state, measured as GFR (determined by the inulin-clearance technique)
GFR | 8 weeks
  Changes from baseline following 8-week treatment on renal hemodynamics in both the fasting and postprandial state, measured as GFR (determined by the inulin-clearance technique)

SECONDARY OUTCOMES:
Renal tubular function | 16 weeks
  24-hour urine sodium-, potassium-, chloride-, calcium-, magnesium-, phosphate-, uric acid-, bicarbonate-, ammonium-, urea- and glucose excretion, urine osmolality and urinary pH
Renal tubular function | 8 weeks
  24-hour urine sodium-, potassium-, chloride-, calcium-, magnesium-, phosphate-, uric acid-, bicarbonate-, ammonium-, urea- and glucose excretion, urine osmolality and urinary pH
Renal Damage | 16 weeks
  24-hour urinary albumin excretion, albumin/creatinine ratio (UCR)
Renal Damage | 10 weeks
  24-hour urinary albumin excretion, albumin/creatinine ratio (UCR)
Renal Damage | 8 weeks
  24-hour urinary albumin excretion, albumin/creatinine ratio (UCR)
Renal Damage | 2 weeks
  24-hour urinary albumin excretion, albumin/creatinine ratio (UCR)
Heart Rate (Dinamap®) | 16 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)
Heart Rate (Dinamap®) | 10 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)
Heart Rate (Dinamap®) | 8 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)
Heart Rate (Dinamap®) | 2 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)
Blood Pressure (Dinamap®) | 16 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)
Blood Pressure (Dinamap®) | 10 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)
Blood Pressure (Dinamap®) | 8 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)
Blood Pressure (Dinamap®) | 2 weeks
  Measured using an automated oscillometric blood pressure device (Dinamap®)

OTHER OUTCOMES:
Body anthropometrics: Body mass index | 16 weeks
  Body mass index
Body anthropometrics: Body mass index | 8 weeks
  Body mass index
Body anthropometrics: Body weight | 16 weeks
  Body weight
Body anthropometrics: Body weight | 8 weeks
  Body weight
Body anthropometrics: Height | 16 weeks
  Height
Body anthropometrics: Height | 8 weeks
  Height
Body anthropometrics: Waist circumference | 16 weeks
  Waist circumference
Body anthropometrics: Waist circumference | 8 weeks
  Waist circumference
Body anthropometrics: Hip circumference | 16 weeks
  Hip circumference
Body anthropometrics: Hip circumference | 8 weeks
  Hip circumference
Body fat content | 16 weeks
  Body fat content by bioimpedance analysis
Body fat content | 8 weeks
  Body fat content by bioimpedance analysis
Blood pressure (NexFin®) | 16 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Blood pressure (NexFin®) | 8 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Heart Rate (NexFin®) | 16 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Heart Rate (NexFin®) | 8 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Stroke Volume | 16 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Stroke Volume | 8 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Cardiac output | 16 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Cardiac output | 8 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Cardiac index | 16 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Cardiac index | 8 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Total systemic vascular resistance | 16 weeks
  Continuous beat-to-beat hemodynamic monitor (NexFin®)
Total systemic vascular resistance | 8 weeks
  Continuous beat-to-beat hemodynamic monitor (NexFin®)
Cardiac autonomic nervous system function | 16 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Cardiac autonomic nervous system function | 8 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Microvascular function | 16 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Microvascular function | 8 weeks
  Measured by continuous beat-to-beat hemodynamic monitor (NexFin®)
Arterial stiffness | 16 weeks
  Assessed by radial artery applanation tonometry (SphygmoCor®)
Arterial stiffness | 8 weeks
  Assessed by radial artery applanation tonometry (SphygmoCor®)
Insulin sensitivity (M-value) | 16 weeks
  Derived from the glucose infusion rate during the euglycemic clamp (M-value)
Insulin sensitivity (M-value) | 8 weeks
  Derived from the glucose infusion rate during the euglycemic clamp (M-value)
Insulin sensitivity (OGIS) | 16 weeks
  Meal tolerance test (OGIS)
Insulin sensitivity (OGIS) | 8 weeks
  Meal tolerance test (OGIS)
Insulin sensitivity (Matsuda index) | 16 weeks
  Meal tolerance test (Matsuda index)
Insulin sensitivity (Matsuda index) | 8 weeks
  Meal tolerance test (Matsuda index)
Beta-cell function (insulinogenic index) | 16 weeks
  Meal tolerance test (insulinogenic index)
Beta-cell function (insulinogenic index) | 8 weeks
  Meal tolerance test (insulinogenic index)
Beta-cell function (HOMA-B) | 16 weeks
  HOMA-B
Beta-cell function (HOMA-B) | 8 weeks
  HOMA-B
Beta-cell function (ratio of postprandial glucose and C-peptide) | 16 weeks
  Meal tolerance test (ratio of postprandial glucose and C-peptide)
Beta-cell function (ratio of postprandial glucose and C-peptide) | 8 weeks
  Meal tolerance test (ratio of postprandial glucose and C-peptide)
Lipid spectrum | 16 weeks
  (triglycerides (TG), total-cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C)
Lipid spectrum | 8 weeks
  (triglycerides (TG), total-cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C)
DPP-4 | 16 weeks
  DPP-4 activity
DPP-4 | 8 weeks
  DPP-4 activity
ACE | 16 weeks
  ACE activity
ACE | 8 weeks
  ACE activity
HbA1c (%) | 16 weeks
  HbA1c (%)
HbA1c (%) | 8 weeks
  HbA1c (%)
Fasting plasma glucose (mmol/L) | 16 weeks
  Fasting plasma glucose (mmol/L)
Fasting plasma glucose (mmol/L) | 8 weeks
  Fasting plasma glucose (mmol/L)
Postprandial plasma glucose (mmol/L) | 16 weeks
  Postprandial plasma glucose (mmol/L)
Postprandial plasma glucose (mmol/L) | 8 weeks
  Postprandial plasma glucose (mmol/L)
Free Fatty Acids (FFA) (mmol/L) | 16 weeks
  Free Fatty Acids (FFA) (mmol/L)
Free Fatty Acids (FFA) (mmol/L) | 8 weeks
  Free Fatty Acids (FFA) (mmol/L)
Insulin (mg/L) | 16 weeks
  Insulin (mg/L)
Insulin (mg/L) | 8 weeks
  Insulin (mg/L)
Glucagon (mg/L) | 16 weeks
  Glucagon (mg/L)
Glucagon (mg/L) | 8 weeks
  Glucagon (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mark HH Kramer, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No